CLINICAL TRIAL: NCT02080676
Title: Effects of Marihuana Use on Optic Nerve Parameters and Ocular Blood Flow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, Professor, Carmel Medical Center
Other Study IDs: CMC-14-0001-CTIL
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Intra Ocular Pressure
Keywords: Cannabis; Intra ocular pressure; Ocular perfusion; Blood pressure
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of study: to check the effect of medical cannabis given for approved medical indications on ocular parameters including intra ocular pressure, optic nerve fibers thickness and choroidal thickness.

DETAILED DESCRIPTION:
Purpose of study: to check the effect of medical cannabis given for approved medical indications on ocular parameters including intra ocular pressure, Retinal Nerve Fiber Layer (RNFL) thickness, optic nerve fibers thickness and choroidal thickness.

Adult patients with no ocular pathology that are being treated in the neurology or pain clinics with medical cannabis for different indications, were examined in the eye clinic.

First examination took place after the patient was not smoking for 5 hours. Three more examinations took place 1 hour 3 hours and 5 hours after smoking cannabis.

The following parameters were checked: blood pressure, pulse, visual acuity, intra ocular pressure, corneal thickness, axial length, slit lamp examination of anterior segment, fundoscopy and Optical Coherence Tomography (OCT) of the retina, and optic nerve.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Treated with medical cannabis for approved medical indications

Exclusion Criteria:

* Known ocular pathology
* Topical or systemic treatment for intra ocular pressure
* Previous topical, intra ocular or systemic steroid treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over the age of 18, with no ocular pathology that are being treated in the neurology or pain clinics with medical cannabis for different indications.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Intra ocular pressure | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel